CLINICAL TRIAL: NCT06637553
Title: Effects of Adlay Extract Formula on Dysmenorrhea in Women
Acronym: ECCEMPW
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Shih-Min Hsia, distinguished professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N201708023
Record Dates: First submitted 2024-10-04; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Dysmucorrhea; Menstrual Pain
Keywords: Dysmenorrhea; Adlay formula
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Same weight as the treatment dissolved in 200cc of hot water once daily for 3 menstrual cycle
  Interventions: Combination Product: Placebo
- Treatment (Experimental): The extract will be administered at a dose of 20 grams dissolved in 200cc of hot water once for 3 menstrual cycledaily
  Interventions: Combination Product: Adlay formula

INTERVENTIONS:
Combination Product: Adlay formula — The extract will be administered at a dose of 20 grams dissolved in 200cc of hot water once daily
  Arms: Treatment
Combination Product: Placebo — Same weight as the adlay formula but did not include the active compound
  Arms: Placebo

SUMMARY:
Due to the Westernization of diet in Taiwan, the risk of many chronic diseases has increased. Some diseases and improper treatments are closely related to menstrual pain and functional impairment in women. Women's menstrual pain can affect daily life and work, and many plant-based extracts have been found to have beneficial effects on alleviating menstrual pain. Therefore, the development of functional health food that can improve menstrual pain is of great significance for health promotion and the market.

Coix seed has long been understood to have properties beneficial for menstrual health. Scientific research has demonstrated its effectiveness in alleviating menstrual pain. The primary ingredient, "coix seed extract," has been extensively studied, and its efficacy has been confirmed through numerous clinical and animal experiments. This study aims to scientifically investigate the effect of coix seed compound extract on menstrual pain in women and to understand its underlying mechanism and potential benefits.

DETAILED DESCRIPTION:
This study investigates the efficacy of coix seed compound extract in alleviating menstrual pain and its potential impact on inflammatory markers. The study will enroll women aged 20-40 with a history of moderate to severe menstrual pain, especially on the first or second day of menstruation. The study includes participants with regular menstrual cycles of 21-35 days.

Participants who meet the inclusion criteria will undergo a series of blood tests throughout the study. Blood samples (10cc each) will be collected three times-once before the intervention, and twice during the treatment period-to assess inflammatory markers, including IL-6 and cytokines. The samples will be analyzed for blood biochemical parameters and stored for future evaluations.

The intervention involves the daily administration of 20 grams of coix seed compound extract dissolved in 200cc of hot water, starting one day before menstruation and continuing for the duration of each menstrual cycle during the study period. The compound includes a mixture of coix seed extract, grape seed extract, and cranberry extract, which are recognized as safe food ingredients.

Potential side effects are expected to be minimal due to the natural composition of the extract. However, participants will be monitored for any adverse reactions. In the event of side effects, participants will be advised to discontinue the extract and consult with the research team.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20-40
* Women who have experienced menstrual pain in recent years, especially on the first or second day of menstruation
* Women whose menstrual pain affects their daily life
* Women with a regular menstrual cycle of 21-35 days, with menstruation lasting 3-7 days

Exclusion Criteria:

* Pregnant or breastfeeding women, or those planning pregnancy or using birth control
* Women with severe gynecological diseases
* Women who have undergone uterine surgery or recent pelvic surgery
* Women with major diseases such as cancer, heart disease, or thyroid disorders
* Women who have used pain relief medication for menstrual pain in the past month

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Dysmenorrhea only in female
Enrollment: 77 (Actual)
Dates: Start 2017-10-14 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Pain relief | Pain levels will be measured at baseline and after each menstrual cycle during the 3-month intervention period
  Pain relief will be assessed using the Visual Analog Scale (VAS), which measures pain intensity on a scale from 0 (no pain) to 10 (worst pain imaginable). Participants will report their pain levels at specific time points.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical Univeersity, Taipei, Xinyi, Taiwan

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available